CLINICAL TRIAL: NCT00253097
Title: The Post Stroke Preventive Trial (PREVENT) A Randomised Controlled Trial Nested in a Cohort (RIALTO) Study
Brief Title: The Post Stroke Preventive Trial (PREVENT). A RCT Nested in a Cohort Study
Acronym: PREVENT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Nete Hornnes Research Director, Ph.d-student, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: KFE 003
Record Dates: First submitted 2005-11-14; First posted 2005-11-15 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-07

CONDITIONS: Cerebrovascular Accident; Transient Ischemic Attack; Myocardial Infarction
Keywords: stroke recurrence; risk factors; health behavior; intervention; tertiary prevention
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Myocardial Infarction; Health Behavior | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Patients in the control group had the usual care provided at the stroke unit, that is counselling on avoiding risky health behavior, compliance with preventive medication, measurement of blood pressure and a 3 months' visit in the outpatient clinic
  Interventions: Behavioral: Intervention
- Intervention (Experimental): Patienta allocated to the intervention group have 4 visits by a study nurse. She will measure patient's blood pressure (BP) by standardized meathods, inform the patient about the target BP, stress the importance of lowering the BP and in case of elevated BP she advices the patient to go the the GP for further control. She advises about smoking cessation, reduction of alcohol consumption, loss of excess body weigt and stresses the importance of physical activity as appropriate
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Patients allocated to the intervention group have 4 visits by a study nurse. She will measure patient's blood pressure (BP) by standardized meathods, inform the patient about the target BP, stress the importance of lowering the BP and in case of elevated BP she advices the patient to go the the GP for further control. She advises about smoking cessation, reduction of alcohol consumption, loss of excess body weigt and stresses the importance of physical activity as appropriate

SUMMARY:
Patients with a diagnosis of stroke or TIA, who are already included in the RIALTO-cohort study are asked to participate in a RCT after discharge from hospital.

Patients in the intervention group will receive four visits by a study nurse with the aim of controlling the patient's hypertension, reducing risk factors like tobacco smoking and obesity, and motivating the patient to physical activity and to a healthy diet.Patients in the control group will receive the usual treatment.

This study is aimed at testing the hypothesis, that

Primary outcome: the blood pressure lowering will be greater in the intervention group Secondary outcomes: the blood pressure will be lower in the intervention group and the number of patients who have stopped smoking will be greater in the intervention group The number of obese patients who have reduced their BMI will be greater in the intervention group The number of patients with a Rankin Scale<3 who are physically active for four hours a week will be greater in the intervention group Time to recurrent stroke, MI and death will be longer in the intervention group

Outcomes are measured by follow up visit one and two years after inclusion in the study

Expected Total Enrollment: 342 in the RCT, 1200 in the cohort

Study Start: 011205 (PREVENT) Study Completion: January 2009(PREVENT), September 2013 (RIALTO Cohort study)

DETAILED DESCRIPTION:
Stroke survivors are at risk of cerebrovascular and cardiovascular complications. In Denmark 25% of stroke admissions are caused by recurrent stroke or TIA. Little is known of the risk factors for recurrent stroke. This is being investigated in a cohort study (RIALTO) initiated in may 2004. The PREVENT study is aimed at studying the health behavior of stroke survivors as well as the effect of a preventive intervention aimed at risk factors associated with hypertension. Hypertension is the main risk factor for primary stroke and the one risk factor known to be associated with stroke recurrence.

Inclusion criteria: inclusion in the RIALTO-cohort, no severe cognitive deficits or dementia, no other life threatening disease.

Exclusion criteria: discharge to a nursing home

Participants (n=342) are randomised to either the intervention group (n=171) or the control group (n=171). Randomisation is performed by a computer-generated allocation schedule, with the randomisation sequence blocked from previewing. The analyser will be blinded from the allocation of the patients.

Baselinedata: Blood pressure, BMI and Rankin scale will be monitored few days prior to discharge.Blood pressure will be measured according to standards set by the Danish Society of hypertension.

Patients in the intervention group will receive a visit by a study nurse one, four, seven, and ten months after discharge. The aim of the visits are: controlling the patient's hypertension, reducing risk factors like tobacco smoking and obesity, motivating the patient to physical activity and to a healthy diet as well as compliance with pharmacological treatment of hypertension, diabetes, hypercholesterolemia and anti-thrombotic treatment.Patients in the control group will receive the usual treatment.

This study is aimed at testing the hypothesis, that

Primary outcome: the blood pressure lowering will be greater in the intervention group Secondary outcomes: the blood pressure will be lower in the intervention group and the number of patients who have stopped smoking will be greater in the intervention group The number of obese patients who have reduced their BMI will be greater in the intervention group The number of patients with a Rankin Scale<3 who are physically active for four hours a week will be greater in the intervention group Time to recurrent stroke, MI and death will be longer in the intervention group

Outcomes are measured by follow up visit one and two years after inclusion in the study. Hypertension is defined as a blood pressure > 140 mm Hg or > 90 mm Hg. The diagnosis of a recurrent stroke will be based on a CT og MR scan or on the clinical diagnosis made by a neurologist.MI should be confirmed by an ECG and by relevant biomarkers.

All participants will be followed up by register data for six years from inclusion as will all participants of the RIALTO cohort.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of stroke or TIA inclusion in the RIALTO cohort no severe cognitive deficits or dementia

Exclusion Criteria:

* discharge to a nursing home

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2005-12; Primary Completion 2009-10 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
blood pressure lowering at 12 and 24 months | November 2006 - october 2009

SECONDARY OUTCOMES:
blood pressure | November 2006 - october 2009
BMI | November 2006 - october 2009
Level of physical activity | November 2006 - october 2009
Time to events:Stroke recurrence, MI and death | November 2006 - october 2009
all assessed 12 and 24 months after inclusion in the study | November 2006 - october 2009
Smoking cessation | november 2006 to october 2009

CONTACTS AND LOCATIONS:
Overall Officials: Nete Hornnes, RN, MPH, Study Director — Clinical Research Unit, Hvidovre Hospital
Locations (2):
- Denmark (2):
  - Bispebjerg Hospital, Copenhagen
  - Frederiksb Hospital, Frederiksberg

REFERENCES:
- [Derived] Hornnes N, Larsen K, Brink-Kjaer T, Boysen G. Specific antismoking advice after stroke. Dan Med J. 2014 Apr;61(4):A4816. PMID 24814592